CLINICAL TRIAL: NCT06125522
Title: TACTIVE-U: AN INTERVENTIONAL SAFETY AND EFFICACY PHASE 1B/2, OPEN-LABEL UMBRELLA STUDY TO INVESTIGATE TOLERABILITY, PK, AND ANTITUMOR ACTIVITY OF VEPDEGESTRANT (ARV-471/PF-07850327), AN ORAL PROTEOLYSIS TARGETING CHIMERA, IN COMBINATION WITH OTHER ANTICANCER TREATMENTS IN PARTICIPANTS AGED 18 AND OLDER WITH ER+ ADVANCED OR METASTATIC BREAST CANCER, SUB-STUDY C (ARV-471 IN COMBINATION WITH SAMURACICLIB)
Brief Title: TACTIVE-U: A Study to Learn About the Study Medicine (Vepdegestrant) When Given With Other Medicines in People With Advanced or Metastatic Breast Cancer. (Sub-Study C)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Arvinas Estrogen Receptor, Inc. (Industry); Carrick Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C4891024; 2023-507125-41-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-10-16; First posted 2023-11-09 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: TACTIVE-U; Umbrella study; PROTAC; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase 1b will use an escalation/de-escalation approach to determine the RP2D of ARV-471 when administered in combination with samuraciclib. The decision to escalate the starting dose level of ARV-471 will be using mTPI-2 decision criteria based on the number of DLT-evaluable participants and the number of DLTs in those participants during the DLT observation period (Cycle 1).
  Phase 2 will further evaluate the preliminary antitumor activity and safety of the combination RP2D.
  In addition, the potential drug-drug interaction (DDI) between ARV-471 and samuraciclib will be evaluated, at the doses selected as recommended dose for expansion (RDE(s)), in a DDI Assessment Cohort(s)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ARV-471 in combination with Samuraciclib (Experimental): ARV-471 administered orally QD continuously and Samuraciclib administered orally QD continuously on 28-day cycles
  Interventions: Drug: vepdegestrant; Drug: Samuraciclib

INTERVENTIONS:
Drug: vepdegestrant — Daily oral dosages of ARV-471 continuously, dose escalation/de-escalation in Phase 1b until RP2D determined, cycles lasting 28 days
  Other Names: ARV-471 / PF-07850327
Drug: Samuraciclib — Daily oral dosages of Samuraciclib continuously, dose escalation/de-escalation in Phase 1b until RP2D determined, cycles lasting 28 days

SUMMARY:
The purpose of this study is to learn about the safety and effects of the study medicine called vepdegestrant. The safety and effects of vepdegestrant will be see when given with other medicines. Vepdegestrant is studied to see if it can be a possible treatment for advanced metastatic breast cancer. This type of cancer would have spread from where it started (breast) to other parts of the body and would be tough to treat.

The study is seeking for participants who have breast cancer that:

* is hard to treat (advanced) and may have spread to other organs (metastatic). is sensitive to hormonal therapy (it is called estrogen receptor positive).
* is no longer responding to treatments taken before starting this study.

This study is divided into separate sub-studies.

For Sub-Study C:

All the participants will receive vepdegestrant and a medicine called samuraciclib.

Vepdegestrant and samuraciclib will be taken once in a day by mouth. The medicines will be taken at home. The experience of people receiving the study medicines will be studied. This will help see if the study medicine is safe and effective.

Participant will continue to take vepdegestrant and samuraciclib until:

* their cancer is no longer responding, or
* side effects become too severe.

They will have visits at the study clinic about every 4 weeks.

DETAILED DESCRIPTION:
C4891024 is a prospective, open-label, multicenter, Phase 1b/2 sub-study to evaluate the safety, antitumor activity, and PK of ARV-471 with samuraciclib in the treatment of participants with A/MBC. The sub-study is part of Umbrella platform, TACTIVE-U, comprising multiple sub-studies that independently evaluate ARV-471 in participants with Estrogen Receptor Positive/Human Epidermal Growth Factor Receptor 2 Negative (ER+/HER2-) Advanced or Metastatic Breast Cancer. ARV-471 will act as the backbone therapy given in combination with other anticancer agents thought to have clinical relevance in ER+ breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of breast cancer. At time of enrollment this must not be amendable to surgical resection with curative intent (≥1% ER+ stained cells as per local practice on the most recent tumor biopsy HER2- tumor by IHC or in-situ hybridization per ASCO/CAP).
* prior anticancer therapies: up to 2 lines of prior therapies for advanced/metastatic disease; 1 line of any CDK4/6 inhibitor-based regimen is required (in any setting eg adjuvant, metastatic)
* at least 1 measurable lesion as defined by RECIST v1.1.
* ECOG PS ≤1.

Exclusion Criteria:

* visceral crisis at risk of life-threatening complications in the short term
* known history of drug-induced pneumonitis or other significant symptomatic deterioration of lung functions.
* newly diagnosed brain metastases, or symptomatic CNS metastases, carcinomatous meningitis, or leptomeningeal disease. Participants with a history of CNS metastases or cord compression are eligible if they have been definitively treated, clinically stable and discontinued anti-seizure medications and corticosteroids for at least 28 days prior to enrollment in the of study.
* history of any other tumor malignancies within the past 3 years, except for the following: (1) adequately treated basal or squamous cell carcinoma of the skin; (2) curatively treated in situ carcinoma of the cervix.
* inflammatory breast cancer
* impaired cardiovascular function or clinically significant cardiovascular diseases
* concurrent administration of medications, food, or herb supplements that are strong inhibitors/inducers of CYP3A, strong CYP2D6 inhibitors and drugs known to predispose to Torsade de Pointes or QT interval prolongation.
* renal impairment, not adequate liver function and/or bone marrow function
* known active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1b: Number of Participants With Dose Limiting Toxicities | 28 days
  Dose Limiting Toxicities rate for ARV-471 in combination with Samuraciclib, estimated based on data from DLT-evaluable participants during the DLT observation period (Cycle 1).
Drug Drug Interaction: To evaluate the effect of samuraciclib on PK of ARV 471. | From the start of Lead-in period (maximum 13 days) to the end of cycle 1 (at least 28 days)
  Steady-state Area under the plasma concentration versus time curve (AUCtau) of ARV-471 with and without coadministration of samuraciclib
Drug Drug Interaction: To evaluate the effect of samuraciclib on PK of ARV 471. | From the start of Lead-in period (maximum 13 days) to the end of cycle 1 (at least 28 days)
  Steady-state Peak Plasma concentration ( Cmax) of ARV-471 with and without coadministration of samuraciclib
Phase 2: Percentage of Participants With Objective Response by investigator assessment | Up to approximately 1 year
  Objective response (OR) refers to confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1. as determined by investigator assessment.
Drug Drug Interaction: • To evaluate the effect of ARV 471 on PK of samuraciclib. | From the start of Lead-in period (maximum 13 days) to the end of cycle 1 (at least 28 days))
  Single dose AUC0-72 of samuraciclib with and without coadministration of ARV 471.
Drug Drug Interaction: • To evaluate the effect of ARV 471 on PK of samuraciclib. | From the start of Lead-in period (maximum 13 days) to the end of cycle 1 (at least 28 days))
  Single dose Cmax of samuraciclib with and without coadministration of ARV 471.

SECONDARY OUTCOMES:
Phase 1b, Drug drug interaction and Phase 2: Evaluation of Safety and Tolerability of ARV-471 in combination with Samuraciclib | First study drug dose through a minimum of 28 Days After Last study drug administration
  AEs as characterized by type, frequency, intensity as graded by NCI CTCAE version 5.0, timing, seriousness, and relationship to ARV-471 in combination with samuraciclib.
  Laboratory test abnormalities as characterized by type, frequency, intensity (as graded by NCI CTCAE version 5.0), and timing.
  Changes from baseline for the ECG parameters heart rate, QTcF, PR interval, and QRS complex will be summarized by treatment and time. The frequency of uncorrected QT values above 500 ms will be tabulated.
Phase 1b: To evaluate antitumor activity of ARV-471 in combination with samuraciclib | Up to approximately 1 year
  Objective response (OR) refers to confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1. as determined by investigator assessment.
Phase 1b and Phase 2: Duration of Response by investigator assessment. | Up to approximately 1 year
  Duration of Response (DoR) is defined for participants with confirmed OR (CR or PR) as the time from the first documentation of OR to the first documentation of objective tumor progression or to death due to any cause, whichever occurs first.
Phase 1b and Phase2: Percentage of participants with Clinical Benefit Response by investigator assessment. | Up to approximately 1 year
  Clinical Benefit Response (CBR) is defined as the proportion of participants with Best Overall Response of confirmed CR or PR at any time, or Stable Disease (SD) ≥24 weeks
Phase 1b and Phase 2: Progression Free Survival by investigator assessment. | Up to approximately 1 year
  Progression Free Survival (PFS) is defined as the time from the date of first dose of study interventions to the date of first documentation of PD or death due to any cause, whichever occurs first.
Phase 1b and Phase 2: Plasma concentrations of ARV-471 and samuraciclib. | At predefined intervals throughout the treatment period, up to cycle 7 (each cycle is 28 days)
  To evaluate the plasma exposure of ARV-471 and samuraciclib when ARV-471 and samuraciclib are given in combination.
Phase 1b: Evaluation of effect of samuraciclib on PK of ARV-471 | At predefined intervals throughout the treatment period, up to cycle 7 (each cycle is 28 days)
  AUCtau of ARV-471 with and without co-administration of samuraciclib
Phase 1b: Evaluation of effect of samuraciclib on PK of ARV-471 | At predefined intervals throughout the treatment period, up to cycle 7 (each cycle is 28 days)
  Cmax of ARV-471 with and without co-administration of samuraciclib
Phase 2:ctDNA plasma quantitative changes from pre-treatment | At predefined intervals throughout the treatment period, up to cycle 3 (each cycle is 28 days) and end of treatment
  To assess changes from baseline levels in plasma ctDNA with treatment and to evaluate potential predictability of their associations with clinical outcomes.
Phase 2: To evaluate the correlation between TP53 mutation status and antitumor activity | Screening
  Participants classified on basis of pathological TP53 mutation detected or not detected.
Phase 2: Overall Survival | Through study completion, up to approximately 3 year
  Overall Survival (OS) is defined as the time from the date of first dose of study interventions to the date of death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (21):
- United States (17):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Highlands Oncology Group, Rogers, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - Clinical and Translational Research Unit (CTRU), Palo Alto, California
  - Stanford Cancer Center, Palo Alto, California
  - UCHealth Poudre Valley Hospital, Fort Collins, Colorado
  - UCHealth Harmony, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth - Medical Center of the Rockies, Loveland, Colorado
  - Memorial Hospital East, Shiloh, Illinois
  - Siteman Cancer Center - Shiloh, Shiloh, Illinois
  - Siteman Cancer Center - St Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Siteman Cancer Center - North County, Florissant, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
- Institut Jules Bordet, Anderlecht, Bruxelles-capitale, Région de, Belgium
- Centre Georges François Leclerc, Dijon, Côte-d'or, France
- Italy (2):
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Lombardy
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore, Roma

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4891024